CLINICAL TRIAL: NCT03841695
Title: The Therapeutic Effect of the Rehabotics Medical Technology Corporation (RMTC) Finger-hand Robot on Upper-limb Rehabilitation of Stroke Patients
Brief Title: The Therapeutic Effect of the Hand Robot on Stroke Patients Upper-lime Rehabilitation of Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201800703A3C601
Record Dates: First submitted 2018-12-20; First posted 2019-02-15 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Experimental group received Robot Assisted Training (RMTC finger-hand robot (Mirror Hand)) and traditional occupation therapy (Conventional OT) for 1 hour and forty minutes.
  Interventions: Device: RMTC finger-hand robot (Mirror Hand); Other: Conventional OT
- Control Group (Active Comparator): Control group received traditional occupation therapy (Conventional OT) for 1 hour and forty minutes.
  Interventions: Other: Conventional OT

INTERVENTIONS:
Device: RMTC finger-hand robot (Mirror Hand) — The robotic hand will apply on the patient's affected hand and the sensor glove will apply on the patient's un-affected hand, the patient can manipulate their affected hand by their un-affected hand and do the task oriented bimanual training.
  Arms: Treatment Group
Other: Conventional OT — The focus of occupational therapy is to help individuals achieve health, well-being, and participation in life through engagement in activities (American Occupational Therapy Association [AOTA], 2014). For stroke rehabilitation, occupational therapy includes retraining in self-care skills, addressing ongoing deficits such as weakness, sensory loss, and cognitive impairments that limit engagement in activities of daily living, and training in community reintegration and modifying tasks or environments.

SUMMARY:
In the present study, the RMTC finger-hand robot and combined with the mechanism of neuroplasticity will be used on the upper-limb rehabilitation of stroke patients. The participants will be randomized assigned to treatment group (TG, robot assisted treatment) and control group (CG, conventional treatment). In the experimental group, task oriented bi-manual training will be applied using the unaffected hand to guide the affected hand by RMTC robot system. The investigators will estimate the motor function of distal part of upper-limb before and after treatments. The results will be compared with the convention rehabilitation treatment. The primary outcomes are Fugl-Meyer assessment (FMA); and the secondary outcome measurements are modified Ashworth scale (MAS),Action Reach Arm Test (ARAT), Box & block test、Brunnstrom recovery Stage, and motor activity log (MAL).

DETAILED DESCRIPTION:
Clinical reports indicated the functional recovery of the distal part of upper limb in stroke patient needs time period longer than other body parts, and there is a limitation in the efficiency of conventional treatment on the distal part of upper limb. Robot assisted rehabilitation is a novel application in treatment. Rehabilitation robot is able to assist patients move the affected side through external power to achieve a repeated exercising and further evoke the motor function. In the present study, the wearable RMTC finger-hand robot and combined with the mechanism of neuroplasticity will be used on the upper-limb rehabilitation of stroke patients. The patient (post stroke>1 month) age from 20-90 years old with Modified Ashworth Scale ≦2, Brunnstrom Recovery Stage of Arm ≧ 2, Mini-Mental State Examination ≧24 will be included as our participation. The participants will be randomized assigned to treatment group (TG, robot assisted treatment, n=30) and control group (CG, conventional treatment, n=30). In the treatment group, task oriented bi-manual training will be applied using the unaffected hand to guide the affected hand by RMTC robot system, the patient will also receive additional conventional treatment. In the control group, the patient will receive 100 minutes conventional treatment. The investigators will estimate the motor function of distal part of upper-limb before and after treatments. The results will be compared with the convention rehabilitation treatment. The primary outcomes are Fugl-Meyer assessment (FMA); and the secondary outcome measurements are modified Ashworth scale (MAS),Action Reach Arm Test (ARAT), Box & block test、Brunnstrom recovery Stage, and motor activity log (MAL). The investigators will follow up the patient at the 3rd and 6th month after complete trial.

ELIGIBILITY:
Inclusion Criteria:

* Modified Ashworth Scale, MAS≦2
* Brunnstrom Recovery Stage of Arm≧2
* Mini-Mental State Examination; MMSE≧24
* aged from 20-90 years
* first stroke ≧1 month

Exclusion Criteria:

* poor cognitive ability (such as moderate to severe dementia, etc.) or mental illness (such as convulsions)
* wrist musculoskeletal system disease (such as fractures, tendon rupture, etc.) can not withstand external forces
* skin disorders (such as pressure sores, trauma, cellulitis, etc.)
* cerebellar stroke

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change of Fugl-Meyer Assessment (FMA-Upper limb) | Measurement will be performed at pre-treatment (0 months), treatment completion (post-treatment, an average of 4 weeks), 1 and 3 months (follow-up)
  Fugl-Meyer assessment is an stroke specific index for estimating the performance of motor function, Total scores of FMA-Upper limb ranged from 0-66.

SECONDARY OUTCOMES:
Change of Modified Ashworth Scale (MAS) | Measurement will be performed at pre-treatment (0 months), treatment completion (post-treatment, an average of 4 weeks), 1 and 3 months (follow-up)
  The MAS is an index for estimating the muscle spasticity, minimal is MAS=0 and maximal is MAS=4.
Change of Action Research Arm Test (ARAT) | Measurement will be performed at pre-treatment (0 months), treatment completion (post-treatment, an average of 4 weeks), 1 and 3 months (follow-up)
  The ARAT is a measurement for evaluating the alteration of upper limb's motor function. Total scores of ARAT ranged from 0-57.
Change of Brunnstrom Recovery Stage (BRS) | Measurement will be performed at pre-treatment (0 months), treatment completion (post-treatment, an average of 4 weeks), 1 and 3 months (follow-up)
  The BRS is a measurement tool for estimating the motor recovery consist of 6 sequential stages.
Change of Box & Block Test (BBT) | Measurement will be performed at pre-treatment (0 months), treatment completion (post-treatment, an average of 4 weeks), 1 and 3 months (follow-up)
  The BBT is a measurement for test the unilateral gross manual dexterity. The number of blocks transferred from one compartment of a box to another in 1-minute is counted.
Change of Motor Activity Log (MAL) | Measurement will be performed at pre-treatment (0 months), treatment completion (post-treatment, an average of 4 weeks), 1 and 3 months (follow-up)
  The MAL is obtained by an interview for stroke patients to assess the use of their affected limb in the daily life, scaled from 0-5.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital at Taoyuan, Taoyuan, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Fugl-Meyer AR. Post-stroke hemiplegia assessment of physical properties. Scand J Rehabil Med Suppl. 1980;7:85-93. No abstract available. PMID 6932734
- [Background] Mathiowetz V, Volland G, Kashman N, Weber K. Adult norms for the Box and Block Test of manual dexterity. Am J Occup Ther. 1985 Jun;39(6):386-91. doi: 10.5014/ajot.39.6.386. PMID 3160243
- [Background] CARROLL D. A QUANTITATIVE TEST OF UPPER EXTREMITY FUNCTION. J Chronic Dis. 1965 May;18:479-91. doi: 10.1016/0021-9681(65)90030-5. No abstract available. PMID 14293031
- [Background] Crow JL, Lincoln NB, Nouri FM, De Weerdt W. The effectiveness of EMG biofeedback in the treatment of arm function after stroke. Int Disabil Stud. 1989 Oct-Dec;11(4):155-60. doi: 10.3109/03790798909166667. PMID 2701823
- [Background] Lyle RC. A performance test for assessment of upper limb function in physical rehabilitation treatment and research. Int J Rehabil Res. 1981;4(4):483-92. doi: 10.1097/00004356-198112000-00001. No abstract available. PMID 7333761